# Assessment of Root Apex Position of Mandibular Molars and Premolars linear to Inferior Alveolar Canal among a sample of Egyptian Population Using CBCT: A Cross sectional study

### **Protocol**

submitted to Faculty of Dentistry, Cairo University for partial fulfillment of the requirements for Master Degree in Oral and Maxillofacial Radiology

Research code:Rad 2:5:1

05/09/2018

Presented by

## Menna Tallah Mosaad El-said

Resident at Oral and Maxillofacial Radiology Department

B.D.S. 2012

Faculty of Dentistry

Cairo University

2018

# **Supervisors**

# Dr. Farid Medhat

Assistant professor of Oral and Maxillofacial Radiology

Faculty of Dentistry

Cairo University

# Dr. Alaa Nawwar

Lecturer of Oral and Maxillofacial Radiology

Faculty of Dentistry

Cairo University

# Introduction

The inferior alveolar nerve (IAN) position is important in avoiding nerve damage during invasive dental procedures. The inferior alveolar bundle is located in the mandibular canal, which runs obliquely through the ramus of the mandible and horizontally through the mandible. The components of the inferior alveolar neurovascular bundle, which is the major supplier of both sensation and blood to the mandible, are arranged consecutively from the superior to inferior positions as follows: vein, artery, and nerve (Yu, Lee, Jeon, Chung, & Kim et al 2016). The IAN, which is a branch of the mandibular nerve ( the third branch of trigmenial nerve), is prone to injury due to trauma, tumors, and a variety of surgical treatments. The IAN provides innervation to the mandibular molars and premolars and their gingiva. The incisive branch, an extension of the IAN, supplies the anterior teeth (Juodzbalys, Wang, & Sabalys et al 2011).

The dental procedures posterior to the mental foramen increases the risk for injuring the IAN as a result of its proximity to the root apices of mandibular premolars and molars (Pogrel et al 2007; Valmaseda et al 2001). The dental procedures may be endodontic procedures (Pogrel et al 2007; Escoda et al 2007), implant placements (Burstein et al 2008; kraut et al 2002), or extraction of mandibular third molar (Valmaseda et al 2001) can cause injury to IAN, or implant placement, resulting in neuropathic pain or partial or complete numbness in the chin area (Microsc et al 2017).

Endodontic therapy might also damage the IAN. Several mechanisms have been proposed, including (1) neurotoxic effect from root canal filling material penetrating the IAN (**Pogrel et al 2007;Valmaseda et al 2001**); (2) mechanical pressure on the nerve caused by overextension of filling material or over

instrumentation with hand or rotary files (**Pogrel et al 2007; Valmaseda et al 2001**); IAN damage has been suggested to occur in 1% of mandibular premolars that receive root canal treatment (**Escoda et al 2007**).

There is an incidence for nerve injury during dental implant placement, resulting from the poor assessment of bone length or excessive length of implant bodies. Therefore to avoid damage of inferior alveolar nerve, it is important to assess the mandibular canal location in the mandible and edentulous space that represent the missing tooth.( **Jui-Ting Hsu et al 2013**)

The nerve injury is unfavorable consequences for the patient (Escoda et al 2007;Burstein et al 2008). If an intimate relation exists, this may have clinical relevance and risk of nerve injury implications in relation to root canal treatment and dental placement of mandibular premolars and molars

# **Rational of the Study**

The linear relation between mandibular premolar and mandibular molars to inferior alveolar canal is not correlated; this study may help to reduce IAN injury during dental and surgical procedures.

# **Statement of the Problem**

Direct nerve damage may be caused by placement of implants, or surgical extraction, or endodontic treatment. All of these may cause temporary or permanent damage to the IAN (poveda et al 2006; Lvovsky et al 2018). These procedure are invasive, and the nerve may be close to the root apex of the posterior teeth. So the clinical relation between inferior alveolar canal and apices of roots of mandibular premolar and molar is important to avoid nerve damage.

# **Review of literature**

#### **List of main databases used in search:**

- Pubmed
- Google Scholar

#### **Keywords:**

- Cone-beam computed tomography- Inferior Alveolar Nerve-Mandibular Premolars- Mandibular Molars -Nerve Injury.

Various dental procedures distal to mental foramen pose a potential iatrogenic cause of inferior alveolar nerve injury (**Escoda et al 2007**), The dental procedures include the surgical and non-surgical procedural, they include the endodontic treatment, implant placement, or extraction of third mandibular molar (**kovisto et al 2011**).

In endodontic treatment obturation, gutta percha is traditionally considered an inert root-filling material, the parasthesia's cases involving gutta percha results from overfill of thermoplastic gutta-percha. If the sealers are excluded from the apices in the mandibular canal space, it can cause nerve injury (**Hiremath et al 2016**).

Injury to the IAN has also been shown with extraction of mandibular third molars (frequency of 1.3%), suggesting that teeth are often close to the nerve. In patients with mental nerve injury, extraction and implant placement have been implicated in 63% of cases with problems (**Kalladka et al 2008**). **Hidenobu et al** reported the relation of third mandibular molar and position of the inferior alveolar nerve without reporting the root apices relation to the nerve.

One of the dentists' objectives is to retain the nature tooth, but if loss of tooth structure, periodontal disease, or trauma is severe, the tooth might be un-restorable. To replace a lost tooth, the treatment option is placement of dental implant to replace the extracted tooth. Immediate implant placement, with apical penetration of the

implant 4–5 mm beyond the previous position of the tooth root into bone for stabilization, can cause injury to the nerve. If the IAN is in close proximity to the root apex of the tooth extracted, implant placement 4–5 mm below the apex of the socket of extracted tooth might cause injury to the nerve. Nerve damage has been reported in 17% of implant cases (**Kubilius et al 2004**). Paresthesia can be as high as 13% in the posterior mandible from implants (**Burstein et al 2008**). Neurosensory problems can be as high as 52% in patients who have received a dental implant (**Kovisto et al 2011**). Although IAN damage is infrequent and the prevalence is not well-defined, it is a serious situation that has unfavorable complication for the patient. Before going procedures with potential for IAN injury, it is critical to determine the location of the inferior alveolar canal with respect to the surrounding structures to avoid injury of anatomical structure (**Burstein et al 2008**).

Jerjes et al 2005 has reported also that the parasthesia of inferior alveolar nerve may result from infection as inflammatory cyst in correspondence with first and second mandibular premolars, while in the mandibular molars, the distance between the root apex and inferior alveolar canal should be in consideration. In the study by Tilotta-Yasukawa et al 2006, the distance of root apex of first mandibular molars from the inferior alveolar nerve varies from 1 and 4 mm and it is less than 1 mm with the second and third mandibular molars. For this reason, the spread of infectious cases to the inferior alveolar nerve that originates from apices of first or second mandibular molar may be quickly involved the nerve even if the periapical lesion size is small(Rachele et al 2016).

In infectious cases, the paresthesia can be the result of a combination of the following mechanisms. (1) Mechanical Pressure: In particular, the expanding infectious process can cause pressure on the nerve fibers. The pressure induces the paresthesia. (2) Microbial Products: in which the products of certain microbes (gram

negative bacteria) can puncture the perineurium with resultant nerve bundle impairment and soiled the conduction.

In view of these potential complications, several studies were conducted to assess the distances between inferior alveolar canal and the root apices of mandibular premolars and molars. However, most studies included only a limited number of specimens (**Kim et al 2010**) or were based on orthogonal and eccentric periapical radiographs or on panoramic radiographs. The value of such analyses is limited because of superimpositions of surrounding structures or distortions (**Bürklein et al 2015**). Although there is too many studies correlate the relation of third molars to inferior alveolar canal ,and also too many studies correlate the relation of molars to the buccal-lingual cortical bone. There is no relation of root apices of the mandibular premolars and molars to the inferior alveolar nerve in a sample of Egyptian population.

Cone-beam computed tomographic (CBCT) imaging provides 3-dimensional (3D) images with a moderate radiation dose (Patel et al 2014), and numerous studies have reported its value in diagnosing spatial relationships between anatomic structures (Temple et al 2016; Tahmasbi et al 2017). So spatial proximity of vital structures such as the inferior alveolar nerve, the incisive canal, and the mental foramen can be accurately assessed and measured (Benavides et al 2012).CBCT can overcome the limitations of radiographs by providing an accurate and 3D image of teeth and surrounding structures. CBCT scans were found to have an error less than that 0.6 % when measuring mandibular anatomy(Ludlow et al 2007). The advantages of CBCT are the weaknesses of 2D intraoral periapical and panoramic radiographic representations. The ability to visualize the area of interest and avoid superimposition permits accurate radiographic interpretation. So it is useful to assess the position of root apex of first and second premolar and mandibular molars to IAN. In other conventional radiographic techniques, there

| al 1996). |
|-----------|

# **Aim of the Study**

The aim of the study is to assess the linear position between the roots of mandibular premolars and molars and the superior border of inferior alveolar canal.

Population: Adults, male and female from Egyptian population

Outcome Variable: Linear measurement of the distance between root apices of

mandibular premolars and molars to the superior border of

IAN.

| | Outcome | <b>Measuring Device</b> | Measuring Unit |
|---|---|---|---|
| | Measured | | |
| | Distance between | | |
| Primary Outcome | root apices of | CBCT software | Millimeters |
| | mandibular | Romexis® | |
| | premolars and | | |
| | molars to inferior | | |
| | alveolar canal | | |

## **Research question:**

Among the mandibular premolars and molars, which roots are the closest to the inferior alveolar canal, in sample of Egyptian Population?

**Materials and Methods** 

**Study Design:** Cross-sectional Study

**Setting and Location:** 

1- The data collection will be obtained from the data base available at Oral &

Maxillofacial Radiology department at faculty of Dentistry, Cairo University.

2- CBCT images will be obtained from Egyptian patients who had CBCT

examination as part of their dental examination, diagnosis or treatment

planning during the years 2018.

**Participants:** 

A total of 162 CBCT scans of mandibular permanent premolars and molars

belonging to Egyptian individuals are selected according to the following:

**Inclusion criteria:** 

First and second mandibular permanent premolars and molars of Egyptian

patients starting from 18 years, males or females.

Intact roots without fractures or cracks.

Posterior teeth are present and their adjacent and opposing teeth.

Absence of radiological evidence of dental malocclusion that could have

altered the position of premolars or molars.

CBCT scans of mandibular first and second premolars and molars using 20

x 10 cm FOV, 0.4mm voxel resolution.

10

#### **Exclusion criteria:**

- Evidence of apicectomy or periapical surgery.
- Odontogenic or non-odontogenic pathology.
- Congenital deformity of the mandible.
- External Root resorption.
- Previous history of fracture of the mandible.
- Tomographic images of poor quality or artifacts interfering with the detection of mandibular canal and apical morphology of the teeth.

#### Variables:

- 1. The crowding and overlapping of the mandibular posterior teeth.
- 2. Extraction of the adjacent or the opposing tooth may cause tilting of the tooth or over eruption of the opposing tooth.
- 3. Attrition of the teeth may cause over eruption of the teeth.
- 4. The presence of dental anamolies may influence the position of the tooth to the inferior alveolar canal.

#### **Data Sources / Measurements:**

Retrospective Data Analysis will be performed after the CBCT images are pooled from the computer database by convenient sampling technique.

CBCT images will be obtained from patients who required CBCT examination as part of their dental examination, diagnosis or treatment planning without exposing them to unnecessary radiation dose for the research purpose.

All the CBCT examinations are scanned by Planmeca Promax 3D<sup>®</sup>, 20 x 10 cm FOV, 0.4 mm voxel resolution, 90 kVp, 8 mA and 13.5 seconds exposure time.

To assess the shortest distance from the root apices to the border of the inferior alveolar canal, the multiplanar reconstruction view of the manufacturer's software viewer (Planmeca Romexis) with its axial, sagittal and coronal plane will be used, and the cross-sectional images through the mandible will be also used.

Cross sectional images will be oriented parallel to the long axis of the tooth, then the shortest distance from the deepest point of root apices and superior border of the inferior alveolar canal will be obtained to be examined (Umut et al 2017).

CBCT images will be interpreted by two oral radiologists independently; blinded from demographic data of the patients and from the results of each other.

All measurements will be assessed, once by the first investigator and then another time two weeks later for intra-observer reliability. The second investigator will assess the measurements once for inter-observer reliability.

Then inter-observational and intra-observational variability between the observers will be evaluated.

#### Bias:

No source of bias.

#### **Study Size:**

The aim of the study is to assess the relationship between the roots of mandibular premolars and molars and the superior border of inferior alveolar canal in Egyptian population. Based on the previous paper by **San Chong, et al,2017**, the prevalence of alveolar nerve 78%. Using a precision of 5, a design effect set at 1 with 95%CI(confidence interval), a total sample size of 162 will be sufficient. The sample size was calculated by Epi info.

Sampling Strategy: The sample will be collected by convenient sampling technique.

#### **Statistical Methods:**

Data will be analyzed using IBM SPSS advanced statistics (Statistical Package for Social Sciences), version 24 (SPSS Inc.,Chicago,IL). Numerical data will be described as mean and standard deviation or median and range. Categorical data will be described as numbers and percantages. Comparsions between male and females for normally distributed numeric variables will be done using Student's ttest while for non-normally distributed numeric variables will be done by Mann-Whitney test. Comparisons between categorical variables will be performed using the chi square test, A p-value less than or equal to 0.05 will be considered statistically significant. All tests will be tailed.

# References

- 1. Aksoy, U., Aksoy, S. and Orhan, K., 2018. A cone-beam computed tomography study of the anatomical relationships between mandibular teeth and the mandibular canal, with a review of the current literature. *Microscopy research and technique*, 81(3), pp.308-314.
- 2. Benavides, E., Rios, H.F., Ganz, S.D., An, C.H., Resnik, R., Reardon, G.T., Feldman, S.J., Mah, J.K., Hatcher, D., Kim, M.J. and Sohn, D.S., 2012. Use of cone beam computed tomography in implant dentistry: the International Congress of Oral Implantologists consensus report. *Implant dentistry*, 21(2).
- 3. Bürklein, S., Grund, C. and Schäfer, E., 2015. Relationship between root apices and the mandibular canal: a cone-beam computed tomographic analysis in a German population. *Journal of endodontics*, 41(10), pp.1696-1700.
- 4. Burstein J, Mastin C, Le B. Avoiding injury to the inferior alveolar nerve by routine use of intraoperative radiographs during implant placement. J Oral Implantol 2008;34:34–8.
- 5. Burstein J, Mastin C, Le B. Avoiding injury to the inferior alveolar nerve by routine use of intraoperative radiographs during implant placement. J Oral Implantol 2008;34:34–8.
- Censi, R., Vavassori, V., Borgonovo, A.E. and Re, D., 2016. Infection Related Inferior Alveolar Nerve Paresthesia in the Lower Premolar Teeth. *Case reports* in dentistry, 2016.
- 7. Claeys V, Wackens G. Bifid mandibular canal: literature review and case report. DentomaxillofacRadiol 2005;34:55–8.

- 8. Escoda-Francoli J, Canalda-Sahli C, Soler A, Figueriredo R, Gay-Escoda C. Inferior alveolar nerve damage because of overextended endodontic material: a problem of sealer cement biocompatibility? J Endod 2007;33:1484–9.
- 9. Hiremath, H., Agarwal, R., Hiremath, V. and Phulambrikar, T., 2016. Evaluation of proximity of mandibular molars and second premolar to inferior alveolar nerve canal among central Indians: A cone-beam computed tomographic retrospective study. *Indian Journal of Dental Research*, 27(3), p.312.
- 10.Hsu, J.T., Fuh, L.J., Tu, M.G., Li, Y.F., Chen, K.T. and Huang, H.L., 2013. The effects of cortical bone thickness and trabecular bone strength on noninvasive measures of the implant primary stability using synthetic bone models. Clinical implant dentistry and related research, 15(2), pp.251-261.
- 11.Jerjes W., Swinson B., Banu B., Al Khawalde M., Hopper C. Paraesthesia of the lip and chin area resolved by endodontic treatment: a case report and review of literature. *British Dental Journal*. 2005;198(12):743–745. doi: 10.1038/sj.bdj.4812412.
- 12. Juodzbalys, G., Wang, H.L. and Sabalys, G., 2011. Injury of the inferior alveolar nerve during implant placement: a literature review. Journal of oral & maxillofacial research, 2(1).
- 13.Kalladka M, Proter N, Benoliel R, Czerninski R, Eliav E. Mental nerve neuropathy:patient characteristics and neurosensory changes. Oral Surg Oral Med Oral Pathol Oral Radiol Endod 2008;106:364–70.
- 14.Kim TS, Caruso JM, Christensen H, Torabinejad M. A comparison of conebeam computed tomography and direct measurement in the examination of the mandibular canal and adjacent structures. J Endod 2010;36:1191–4.
- 15. Kovisto, T., Ahmad, M. and Bowles, W.R., 2011. Proximity of the mandibular canal to the tooth apex. *Journal of endodontics*, *37*(3), pp.311-315.

- 16.Kraut R, Chahal O. Management of patients with trigeminal nerve injuries after mandibular implant placement. J Am Dent Assoc 2002;133:1351–4.
- 17. Kubilius R, Sabalys G, Juodzbalys G, Gedrimas V. Traumatic damage to the inferior alveolar nerve sustained in course of dental implantation. possibility of prevention. Stomatologija, Baltic Dental and Maxillofacial Journal 2004;6:106–10.
- 18.Lazzerini F, Minorati D, Nessi R, Gagliani M, Uslenghi CM. The measurement parameters in dental radiography: A comparison between traditional and digital technics. Radiol Med 1996;91:364-9.
- 19.Ludlow JB, Laster WS, See M, Bailey LJ, Hershey HG (2007)Accuracy of measurements of mandibular anatomy in cone beam computed tomography images. Oral Surg Oral Med Oral Pathol Oral Radiol Endod 103:534–542.
- 20.Lvovsky A, Bachrach S, Kim HC, Pawar A, Levinzon O, Itzhak JB, Solomonov M. Relationship between Root Apices and the Mandibular Canal: A Cone-beam Computed Tomographic Comparison of 3 Populations. Journal of endodontics. 2018 Feb 6.
- 21. Maegawa, H., Sano, K., Kitagawa, Y., Ogasawara, T., Miyauchi, K., Sekine, J. and Inokuchi, T., 2003. Preoperative assessment of the relationship between the mandibular third molar and the mandibular canal by axial computed tomography with coronal and sagittal reconstruction. *Oral Surgery, Oral Medicine, Oral Pathology, Oral Radiology and Endodontics*, 96(5), pp.639-646.
- 22.Microsc Res Tech. 2017;1–7. wileyonlinelibrary.com/journal/jemt VC 2017Wiley Periodicals, Inc. | 1Received: 16 September 2017 | Revised: 19 November 2017 | Accepted: 10 December 2017 DOI: 10.1002/jemt.22980.
- 23. Patel S, Durack C, Abella F, et al. European society of endodontology position statement: The use of CBCT in endodontics. Int Endod J 2014;47:502–4.

- 24.Pogrel MA. Damage to the inferior alveolar nerve as the result of root canal therapy. J Am Dent Assoc 2007;138:65–9.
- 25.Poveda R, Bagan JV, Fernandez JM, Sanchis JM. Mental nerve paresthesia associated with endodontic paste within the mandibular canal: report of a case. Oral Surg Oral Med Oral Pathol Oral Radiol Endod 2006;102:46–9.
- 26.San Chong, B., Gohil, K., Pawar, R. and Makdissi, J., 2017. Anatomical relationship between mental foramen, mandibular teeth and risk of nerve injury with endodontic treatment. Clinical oral investigations, 21(1), pp.381-387.
- 27. Shin, Y., Roh, B.D., Kim, Y., Kim, T. and Kim, H., 2016. Accidental injury of the inferior alveolar nerve due to the extrusion of calcium hydroxide in endodontic treatment: a case report. *Restorative dentistry & endodontics*, 41(1), pp.63-67
- 28. Tahmasbi M, Jalali P, Nair MK, et al. Prevalence of middle mesial canals and isthmi in the mesial root of mandibular molars: an in vivo cone-beam computed tomographic study. J Endod 2017;43:1080–3.
- 29.Temple KE, Schoolfield J, Noujeim ME, et al. A cone beam computed tomography(CBCT) study of buccal plate thickness of the maxillary and mandibular posterior dentition. Clinical Oral Implants Res 2016;27:1072–8.
- 30. Tilotta-Yasukawa F., Millot S., El Haddioui A., Bravetti P., Gaudy J.-F. Labiomandibular paresthesia caused by endodontic treatment: An Anatomic and Clinical Study. *Oral Surgery, Oral Medicine, Oral Pathology, Oral Radiology and Endodontology*. 2006;102(4):e47–e59. doi: 10.1016/j.tripleo.2006.02.017
- 31. Valmaseda-Castellon E, Berini-Aytes L, Gay-Escoda C. Inferior alveolar nerve damage after lower third molar surgical extraction: a prospective study of 1117 surgical extractions. Oral Surg Oral Med Oral Pathol Oral Radiol Endod 2001;92:377–83.

32.Yu, S.K., Lee, M.H., Jeon, Y.H., Chung, Y.Y. and Kim, H.J., 2016. Anatomical configuration of the inferior alveolar neurovascular bundle: a histomorphometric analysis. Surgical and Radiologic Anatomy, 38(2), pp.195-201.